CLINICAL TRIAL: NCT06421324
Title: Interventional Study Focused on Providing Personalised Health Recommendations to the General Population Through an Integrated AI Guided App as a Strategy for Gastric Cancer Prevention (AIDA)
Brief Title: Personalised Health Recommendations to the General Population Through an Integrated AI Guided
Acronym: AIDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIDA_HE
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer; Cancer Prevention; Helicobacter Pylori Infection; Artificial Intelligence
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: In practice, for rare diseases we chose a sample size that will allow estimation of sensitivity of the risk score to a pre-specified precision. We have chosen the sample size assuming that the resulting precancer detection model will have a sensitivity of at least 85%, and so that the lower 95% confidence interval will exceed 76%, with 80% power. The R package MKmisc estimates sample size for a proportion based on the Binomial distribution rather than a Normal approximation. In this case, we have estimated a sample size of 141 GIM + cancer and 141 GIM controls (282 in total). With 5% of samples assumed to be failing to be analysed due to a variety of technical reasons, we would need ~300 samples in total. In addition, to train the system 150 gastric cancer cases will be recruited which will provide pathology samples images and endoscopy images that will be taken as part of the clinical practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy controls (No Intervention): Subjects will be recruited prospectively from the Digestive Medicine/Endoscopy Departments of the centres involved. Patients will be treated according to the medical and patient decisions according to the clinical practice protocols of each site. Sample collection will be performed during a gastroscopy for pathological and molecular characterisation. This gastroscopy will be always indicated within usual clinical practice, so no additional risk is planned for the subjects included.
  Inclusion criteria: Subjects ≥18 years old to whom an endoscopy is performed due to gastric symptoms, without previous history of gastric chronic inflammation or Helicobacter pylori infection
- Gastric cancer controls (No Intervention): Subjects will be recruited prospectively from the Digestive Medicine/Endoscopy Departments of the centres involved. Patients will be treated according to the medical and patient decisions according to the clinical practice protocols of each site. Sample collection will be performed during a gastroscopy for pathological and molecular characterisation. This gastroscopy will be always indicated within usual clinical practice, so no additional risk is planned for the subjects included.
  Inclusion criteria: Subjects ≥18 years old with a diagnosis of Gastric Cancer, to whom a gastroscopy is indicated within clinical care naive for chemotherapy.
- GIM cases (Experimental): Subjects will be recruited prospectively from the Digestive Medicine/Endoscopy Departments of the centres involved. Patients will be treated according to the medical and patient decisions according to the clinical practice protocols of each site. Sample collection will be performed during a gastroscopy for pathological and molecular characterisation. This gastroscopy will be always indicated within usual clinical practice, so no additional risk is planned for the subjects included.
  Inclusion criteria: Subjects ≥18 years old with a diagnosis of GIM or previous or current H. pylori infection, to whom a gastroscopy is indicated within clinical care
  Interventions: Behavioral: Health reccommendations

INTERVENTIONS:
Behavioral: Health reccommendations — Patients are given recommendations according to their risk group, based on the model which already predicted health indicators. This information will be sent to the patient's treating physician so that treatment and recommendations are aligned with the clinical care practice based on the European Code of Cancer guidelines, the H. pylori best practices guidelines and European GIM guidelines
  Arms: GIM cases

SUMMARY:
This clinical study aims to be used to implement and validate the AIDA tool in two phases:

* Phase 1: Risk stratification and personalised recommendations & Model development
* Phase 2: Mechanistic Model (Bioresource) development & testing

DETAILED DESCRIPTION:
The AIDA objective (project) is to develop and validate a multidisciplinary AI-powered assistant that helps clinicians diagnose precancerous inflammation, suggests personalised therapeutic strategies for medical treatment and follow-up, and makes personalised recommendations for monitoring patient health status, thus contributing to gastric cancer prevention. This prospective clinical study aims to implement and validate such tool.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years old with a diagnosis of GIM or previous or current H. pylori infection, to whom a gastroscopy is indicated within clinical care
* Availability of a signed informed consent form to participate in the study

Exclusion Criteria:

* Patients to whom an endoscopy is performed for the follow-up of another illness such as oesophageal varices and/or for therapy such as endoscopic dilation, feeding tube placement or endoscopic resection
* Subjects with a clinical diagnosis of gastric diseases other than GIM or GC
* Patients who have received antimicrobials during the four weeks prior to the endoscopy
* Patients who have received proton pump inhibitors and/or bismuth-based treatments at least two weeks prior to the endoscopy
* Subjects for whom clinical data are not available: H. pylori status, eradication treatment, sex, age, tobacco smoking, and first-degree family history of gastric cancer
* Subjects who lack the mental capacity to understand the nature and requirements of the study and who lack the ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of developing Gastric Cancer based on medical records | At the recruitment stage
  Scoring patients as low (>30) / medium / high risk (<6) according to:
  * Degree of 'healthiness' of lifestyle (1 to 10, with 10 as very low and 10 as very high)
  * Co-morbidities (Yes = 1 / No = 5)
  * H. pylori infection history (Yes = 1 / No = 5)
  * Previous gastric intestinal metaplasia (Yes = 1 / No = 5)
  * Dysplasia or atrophy related to chronic gastritis (Yes = 1 / No = 5)
  * Family history of cancer (Yes = 1 / No = 5)
H. pylori Eradication Therapy Recommendation | From 30 days after the H.Pylori positive test result to one year after the first recommendation
  AI driven H. pylori Eradication Therapy Recommendation
GIM risk score assessment using imaging modalities | At the recruitment stage
  AI driven GIM risk score assessment of pre-cancerous lesions using imaging modalities based on: QLQ C30 and STO22 EORTC questionnaire, Healthy lifestyle questionnaire (adapted from EPICs), Baseline clinical data, If H. pylori positive: adherence to treatment: yes/no; eradication yes/no, If GIM: adherence to follow-up guidelines yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Tania Fleitas, MD, PhD, Principal Investigator — Fundación para la Investigación del Hospital Clínico de Valencia
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website — https://www.aidaeuproject.org/

DOCUMENTS (1):
  • Informed Consent Form (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT06421324/ICF_000.pdf